CLINICAL TRIAL: NCT00152971
Title: A Phase III, Randomized, Parallel-group, Double-blind, Active Controlled Study to Investigate the Efficacy and Safety of Two Different Dose Regimens (75mg Day 1 Followed by 150 mg Day 2-completion, and 110 mg Day 1 Followed by 220 mg Day 2-completion) of Dabigatran Etexilate Administered Orally (Capsules), Compared to Enoxaparin 30 mg Twice a Day Subcutaneous for 12 - 15 Days in Prevention of Venous Thromboembolism in Patients With Primary Elective Total Knee Replacement Surgery
Brief Title: Dabigatran Etexilate vs Enoxaparin in Prevention of Venous Thromboembolism (VTE) Post Total Knee Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1160.24
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Arthroplasty, Replacement, Knee; Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — Enoxaparin

ARMS (3):
- Dabigatran Dose 1 (Experimental): low dose regimen taken once daily
  Interventions: Drug: Dabigatran Dose 1 - day 2 to completion; Drug: Dabigatran Dose 1 - day 1
- Dabigatran Dose 2 (Experimental): high dose regimen taken once daily
  Interventions: Drug: Dabigatran Dose 2 - day 2 to completion; Drug: Dabigatran Dose 2 - day 1
- Enoxaparin (Active Comparator): 30 mg subcutaneously twice daily
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Dabigatran Dose 1 - day 2 to completion — low dose regimen taken once daily
  Arms: Dabigatran Dose 1
Drug: Dabigatran Dose 1 - day 1 — low dose regimen taken once daily
  Arms: Dabigatran Dose 1
Drug: Dabigatran Dose 2 - day 2 to completion — high dose regimen taken once daily
  Arms: Dabigatran Dose 2
Drug: Dabigatran Dose 2 - day 1 — high dose regimen taken once daily
  Arms: Dabigatran Dose 2
Drug: Enoxaparin — 30 mg subcutaneously twice daily
  Arms: Enoxaparin

SUMMARY:
To determine the comparative efficacy and safety of two different doses (75mg day 1 followed by 150 mg day 2-completion, and 110 mg day 1 followed by 220 mg day 2-completion) of dabigatran administered orally (capsules), compared to enoxaparin 30 mg twice a day subcutaneous, in prevention of venous thromboembolism in patients with primary elective total knee replacement surgery

ELIGIBILITY:
Inclusion criteria INCLUSION CRITERIA

1. Patients scheduled to undergo a primary, unilateral elective total knee repla cement.
2. Male or female 18 years of age or older.
3. Patients weighing at least 40 kg.
4. Written informed consent prior to the start of study participation.

Exclusion criteria EXCLUSION CRITERIA

1. History of bleeding diathesis.
2. Constitutional or acquired coagulation disorders that in the investigator's judgment puts the patient at excessive risk for bleeding.
3. Major surgery or trauma (e.g. hip fracture) within the last 3 months.
4. Recent unstable cardiovascular disease, such as uncontrolled hypertension at the time of enrollment (investigator's judgment) or history of myocardial infarction within the last 3 months.
5. Spinal or epidural anesthesia, for which more than 3 attempts (sticks) at placement were made, or the placement was traumatic.

   Please note that patients, who are not excluded under this criterion, are to have the catheter pulled at the completion of surgery.
6. Any history of hemorrhagic stroke or any of the following intracranial pathologies: bleeding, neoplasm, arteriovenous (AV) malformation or aneurysm.
7. History of VTE or pre-existing condition requiring anticoagulant therapy.
8. Clinically relevant bleeding (e.g. gastrointestinal, pulmonary, intraocular or urogenital bleeding) within the last 6 months.
9. Gastric or duodenal ulcer within the last 6 months.
10. Liver disease expected to have any potential impact on survival (e.g. hepatitis B or C, cirrhosis, but not Gilbert's syndrome or hepatitis A with complete recovery).
11. Elevated AST or ALT >2x upper limit of normal, based on central lab results or local lab results within 1 month before enrollment.
12. Known severe renal insufficiency (CrCl < 30 mL/min). In order to determine patient inclusion/exclusion, creatinine clearance (CrCl) needs to be calculated only if serum creatinine is elevated or renal insufficiency is suspected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2615 (Actual)
Dates: Start 2004-11; Primary Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (94):
- United States (59):
  - 1160.24.01074 Capstone Clinical Trials, Inc., Birmingham, Alabama
  - 1160.24.01079 West AL Research, Inc, Northport, Alabama
  - 1160.24.01047 Tucson Orhtopaedic Institute, Tucson, Arizona
  - 1160.24.01025 Martin, Bowen, Hefley Knee and Sports, Little Rock, Arkansas
  - 1160.24.01053 OrthoArkansas, PA, Little Rock, Arkansas
  - 1160.24.01085 Martin, Bowen, Hefley Knee and Sports, Little Rock, Arkansas
  - 1160.24.01041 Core Orthopedic Medical Center, Encinitas, California
  - 1160.24.01034 Glendale Adventist Medical Center, Glendale, California
  - 1160.24.01005 Scripps Clinical Ctr for Orthopedic Rsrch & Educ, La Jolla, California
  - 1160.24.01077 Long Beach VA Healthcare system, Long Beach, California
  - 1160.24.01064 Orthopedic Specialty Institute, Orange, California
  - 1160.24.01031 Colorodo Orthopedic Consultants, PC, Aurora, Colorado
  - 1160.24.01027 Advanced Orthopedic and Sports Medicine Specialists, PC, Denver, Colorado
  - 1160.24.01023 Orthopedic Physicians of Colorado, PC, Engelwood, Colorado
  - 1160.24.01020 Bay Pines VA Medical Center, Bay Pines, Florida
  - 1160.24.01024 Pulmonary Associates of Brandon Clinical Research, Brandon, Florida
  - 1160.24.01030 Alliance Research, Inc., Clearwater, Florida
  - 1160.24.01039 Florida Orthopedic Associates, DeLand, Florida
  - 1160.24.01036 Orthopaedic Associates of South Broward, PA, Hollywood, Florida
  - 1160.24.01010 MIMA Century Research Associates, Melbourne, Florida
  - 1160.24.01062 Miami Institute for Joint Reconstruction, Miami, Florida
  - 1160.24.01040 Southern Clinical Research Consultants, Orlando, Florida
  - 1160.24.01067 Baptist Clinical Research, Pensacola, Florida
  - 1160.24.01001 Boehringer Ingelheim Investigational Site, Pinellas Park, Florida
  - 1160.24.01017 Boehringer Ingelheim Investigational Site, Pinellas Park, Florida
  - 1160.24.01019 Boehringer Ingelheim Investigational Site, Pinellas Park, Florida
  - 1160.24.01029 Coastal Medical Research, Port Orange, Florida
  - 1160.24.01038 James A. Haley VA Hospital, Tampa, Florida
  - 1160.24.01063 Resurgens Orthopaedics, Atlanta, Georgia
  - 1160.24.01072 Resurgeons Orthopedics, Atlanta, Georgia
  - 1160.24.01056 Southern Orthopaedic Specialists, Lawrencville, Georgia
  - 1160.24.01028 Intermountain Research Center, Boise, Idaho
  - 1160.24.01022 Iowa Orthopedic Clinic, Des Moines, Iowa
  - 1160.24.01008 Bluegrass Orthopedic/Musculoskeletal Research, LLC, Lexington, Kentucky
  - 1160.24.01070 Sinai Hospital of Baltimore, Baltimore, Maryland
  - 1160.24.01007 Ortho Associates, Towson, Maryland
  - 1160.24.01059 Rockhill Orthopaedics, Kansas City, Missouri
  - 1160.24.01042 Center for Joint Care, Missoula, Montana
  - 1160.24.01014 Charlotte Orthopedic Specialists, Charlotte, North Carolina
  - 1160.24.01035 Wellington Orthopedics and Sports Medicine, Cincinnati, Ohio
  - 1160.24.01006 VA Medical Center, Oklahoma City, Oklahoma
  - 1160.24.01044 Tulsa Bone and Joint Associates, Tulsa, Oklahoma
  - 1160.24.01002 The Orthopedic and Neurological Center of the Cascades, Bend, Oregon
  - 1160.24.01046 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1160.24.01016, Charleston, South Carolina
  - 1160.24.01073 Coastal Orthopedic Associates, PA, Conway, South Carolina
  - 1160.24.01032 Seton Medical Center, Austin, Texas
  - 1160.24.01003 Texas Orthopedic Associates, Dallas, Texas
  - 1160.24.01090 VA Medical Center, Dallas, Texas
  - 1160.24.01026 James Muntz, MD, Houston, Texas
  - 1160.24.01033 Bone and Joint Clinic of Houston, Houston, Texas
  - 1160.24.01076 Discovery Alliance, Houston, Texas
  - 1160.24.01018 Gill Research Center, Lubbock, Texas
  - 1160.24.01069 Correspondence and Pateint vists, Plano, Texas
  - 1160.24.01015 Unlimited Research, LP, San Antonio, Texas
  - 1160.24.01012 Anderson Orthopedic Clinic, Alexandria, Virginia
  - 1160.24.01052 Swedish Medical Center, Seattle, Washington
  - 1160.24.01057 Orthopedic Specialty Clinic of Spokane, PLLC, Spokane, Washington
  - 1160.24.01082 MultiCare Health System, Tacoma, Washington
- Canada (32):
  - 1160.24.02031 University of Alberta Hospital, Edmonton, Alberta
  - 1160.24.02036 2B2.37 Walter Mackenizie Centre, Edmonton, Alberta
  - 1160.24.02024 Red Deer Regional Hospital, Red Deer, Alberta
  - 1160.24.02032 Kelowna General Hospital, Kelowna, British Columbia
  - 1160.24.02034 Hematology/Oncology Research, Vancouver, British Columbia
  - 1160.24.02025 Grace General Hospital, Winnipeg, Manitoba
  - 1160.24.02007 Orthopaedics 4NE, Fredericton, New Brunswick
  - 1160.24.02027 Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - 1160.24.02021 Rouge Valley Health System, Ajax, Ontario
  - 1160.24.02008 Orthopaedic Surgery, Barrie, Ontario
  - 1160.24.02016 Orthopaedic Surgery, Brantford, Ontario
  - 1160.24.02010 Joseph Brant Memorial Hospital, Burlington, Ontario
  - 1160.24.02001 73 Delhi Street, Guelph, Ontario
  - 1160.24.02014 565 Sanatorium Road, Hamilton, Ontario
  - 1160.24.02004 Grand River Hospital, Kitchener, Ontario
  - 1160.24.02028 NHS- Greater Niagara General Site, Niagara Falls, Ontario
  - 1160.24.02022 Lakeridge Health Oshawa, Oshawa, Ontario
  - 1160.24.02017 1053 Carling Avenue, Ottawa, Ontario
  - 1160.24.02026 Ottawa Hospital - General Campus, Ottawa, Ontario
  - 1160.24.02015 York Central Hospital Research, Richmond Hill, Ontario
  - 1160.24.02029 Niagara Health System St. Catharine's General Site, Saint Catherine's, Ontario
  - 1160.24.02009 2863 Ellesmere Road, Scarborough Village, Ontario
  - 1160.24.02003 46 General Hospital Drive, Stratford, Ontario
  - 1160.24.02033 Thunder Bay Regional Hospital, Thunder Bay, Ontario
  - 1160.24.02002 Toronto East General Hospital Fracture Clinic, Toronto, Ontario
  - 1160.24.02023 North York General Hospital, Toronto, Ontario
  - 1160.24.02030 St. Joseph's Health Centre, Toronto, Ontario
  - 1160.24.02006 206-477 King Street, Welland, Ontario
  - 1160.24.02035 Humber River Regional Hospital, Weston, Ontario
  - 1160.24.02011 Windsor Regional Hospital, Windsor, Ontario
  - 1160.24.02012 Hotel Dieu Grace Hospital, Windsor, Ontario
  - 1160.24.02013 Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
- Mexico (2):
  - 1160.24.05009 Traumatologia, Planta Baja, Guadalajara, Jalisco
  - 1160.24.05004, México
- 1160.24.44001 Ravenscourt Park Hospital, London, United Kingdom

REFERENCES:
- [Derived] Rosencher N, Noack H, Feuring M, Clemens A, Friedman RJ, Eriksson BI. Type of anaesthesia and the safety and efficacy of thromboprophylaxis with enoxaparin or dabigatran etexilate in major orthopaedic surgery: pooled analysis of three randomized controlled trials. Thromb J. 2012 Jun 18;10(1):9. doi: 10.1186/1477-9560-10-9. PMID 22709460

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The treatment period is from first administration of study medication, until 3 days after last administration of study medication. Treatment duration is planned for 12 - 15 days. The study period is from first administration of study medication until day 84 - 91.
Pre-assignment Details: Whilst 2615 patients were enrolled/randomised to treatment post surgery in this trial, only 2596 started treatment. Therefore, 19 patients were randomised but not treated (treatment was planned to start post surgery).
Groups:
- Dabigatran 220mg; Dabigatran 150mg: qd (once daily) oral
- Enoxaparin: 30mg bid (twice daily) subcutaneous
Period: Overall Study
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Started | 857 | 871 | 868
Completed | 806 (Non-completers in 'overall study' table may have completed treatment but not study, and vice versa) | 823 (Non-completers in 'overall study' table may have completed treatment but not study, and vice versa) | 819 (Non-completers in 'overall study' table may have completed treatment but not study, and vice versa)
Not Completed | 51 | 48 | 49
Not completed — Adverse Event | 12 | 10 | 9
Not completed — Protocol Violation | 10 | 11 | 8
Not completed — Lost to Follow-up | 17 | 14 | 13
Not completed — Withdrawal by Subject | 9 | 8 | 14
Not completed — Other | 3 | 5 | 5
Period: Treatment
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Started | 857 | 871 | 868
Completed | 786 (Non-completers in 'treatment' table may have completed study but not treatment, and vice versa) | 808 (Non-completers in 'treatment' table may have completed study but not treatment, and vice versa) | 788 (Non-completers in 'treatment' table may have completed study but not treatment, and vice versa)
Not Completed | 71 | 63 | 80
Not completed — Adverse Event | 49 | 40 | 54
Not completed — Protocol Violation | 8 | 6 | 10
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 5
Not completed — Other | 9 | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin | Total
Number analyzed (Participants) | 857 | 871 | 868 | 2596
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (9.5) | 65.9 (9.5) | 66.3 (9.6) | 66.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 486 | 507 | 504 | 1497
  Male | 371 | 364 | 364 | 1099
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (6.0) | 31.4 (6.1) | 31.4 (6.0) | 31.5 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Venous Thromboembolic Event and All-cause Mortality During Treatment Period
Description: Total Venous Thromboembolic Event (VTE) includes both proximal and distal deep vein thrombosis (DVT) (detected by routine bilateral venography), symptomatic DVT (confirmed by venous compression ultrasound, venography or autopsy) and pulmonary embolism (PE) (confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy).
  All of these components and all deaths were centrally adjudicated by the VTE events committee, which was not aware of the treatment allocation of the patients.
Time Frame: First administration until 12-15 days
Population: Full Analysis Set (all patients who had surgery and were randomised, received treatment, had an evaluable venogram for distal and proximal Deep Vein Thrombosis, or had confirmed symptomatic Deep Vein Thrombosis, Pulmonary Embolism, or had died)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 604 | 649 | 643
Participants | 188 | 219 | 163
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Non-Inferiority or Equivalence — Non-inferiority Analysis with NI margin 9.2% on the absolute risk difference scale; p = 0.0234, Normal approximation — Hierarchical testing procedure: first non-inferiority, second superiority; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 5.8, 95% CI [0.8 to 10.8]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Non-Inferiority or Equivalence — Non-inferiority Analysis with NI margin 9.2% on the absolute risk difference scale; p = 0.0009, Normal approximation — Hierarchical testing procedure: first non-inferiority, second superiority; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 8.4, 95% CI [3.4 to 13.3]

2. Secondary Outcome: Number of Participants With Major Venous Thromboembolic Event and Venous Thromboembolic Event-related Mortality During Treatment Period
Description: Major Venous Thromboembolic Event (VTE) is defined as proximal DVT and PE, as adjudicated by the VTE events committee
Time Frame: First administration until 12-15 days
Population: Full Analysis Set - major (all patients who had surgery and were randomised, received treatment, had an evaluable venogram for proximal Deep Vein Thrombosis, or had confirmed symptomatic Deep Vein Thrombosis, Pulmonary Embolism, or had died by a Venous Thromboembolic Event-related death)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 618 | 656 | 668
Participants | 21 | 20 | 15
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.2139, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 1.2, 95% CI [-0.7 to 3.0]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.3628, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 0.8, 95% CI [-0.9 to 2.5]

3. Secondary Outcome: Number of Participants With Proximal Deep Vein Thrombosis During Treatment Period
Description: Proximal Deep Vein Thrombosis as adjudicated by the VTE events committee
Time Frame: First administration until 12-15 days
Population: Full Analysis Set - pDVT (all patients who had surgery and were randomised, received treatment, had an evaluable venogram for proximal Deep Vein Thrombosis, or had confirmed symptomatic Deep Vein Thrombosis)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 614 | 656 | 664
Participants | 15 | 20 | 10
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.2309, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 0.9, 95% CI [-0.6 to 2.5]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.0602, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 1.5, 95% CI [-0.1 to 3.2]

4. Secondary Outcome: Number of Participants With Total Deep Vein Thrombosis During Treatment Period
Description: Total Deep Vein Thrombosis as adjudicated by the VTE events committee
Time Frame: First administration until 12-15 days
Population: Full Analysis Set - tDVT (all patients who had surgery and were randomised, received treatment, had an evaluable venogram, or had confirmed symptomatic Deep Vein Thrombosis)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 600 | 648 | 639
Participants | 184 | 218 | 158
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.0194, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 5.9, 95% CI [1.0 to 10.9]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.0004, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 8.9, 95% CI [4.0 to 13.9]

5. Secondary Outcome: Number of Participants With Symptomatic Deep Vein Thrombosis During Treatment Period
Description: Symptomatic Deep Vein Thrombosis, confirmed by venous compression ultrasound, venography or autopsy, and as adjudicated by the VTE events committee
Time Frame: First administration until 12-15 days
Population: Full Analysis Set - op (all patients who are treated and operated)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 857 | 871 | 868
Participants | 7 | 6 | 5
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.5774, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 1.0000, Fisher Exact

6. Secondary Outcome: Number of Participants With Pulmonary Embolism During Treatment Period
Description: Pulmonary embolism confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy, and as adjudicated by the VTE events committee
Time Frame: First administration until 12-15 days
Population: Full Analysis Set - op
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 857 | 871 | 868
Participants | 6 | 0 | 5
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.7724, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.0308, Fisher Exact

7. Secondary Outcome: Number of Participants Who Died During Treatment Period
Description: All cause death, as adjudicated by the VTE events committee
Time Frame: First administration until 12-15 days
Population: Full Analysis Set - op
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 857 | 871 | 868
Participants | 1 | 1 | 0
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.4968, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 1.0000, Fisher Exact

8. Secondary Outcome: Number of Participants With Total Venous Thromboembolic Event (VTE) and All-cause Mortality During the Follow-up Period
Description: Total Venous Thromboembolic Event (VTE) includes both proximal and distal deep vein thrombosis (DVT) (detected by routine bilateral venography), symptomatic DVT (confirmed by venous compression ultrasound, venography or autopsy) and pulmonary embolism (PE) (confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy).
Time Frame: 3 months
Population: Patients with any data available during follow-up
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 840 | 861 | 853
Participants
  Total VTE and all-cause mortality | 7 | 7 | 10
  asymptotic Deep Vein Thrombosis | 2 | 1 | 4
  symptotic Deep Vein Thrombosis | 2 | 4 | 2
  Pulmonary Embolism | 2 | 0 | 2
  death | 1 | 2 | 2

9. Secondary Outcome: Number of Participants With Bleeding Events (Defined According to Modified McMaster Criteria) During Treatment Period
Description: Major bleeding events were defined as
  * fatal
  * clinically overt associated with loss of haemoglobin >=20g/L in excess of what was expected
  * clinically overt leading to the transfusion of >=2 units packed cells or whole blood in excess of what was expected
  * symptomatic retroperitoneal, intracranial, intraocular or intraspinal
  * requiring treatment cessation
  * leading to re-operation
  Clinically-relevant was defined as
  * spontaneous skin hematoma greater than or equal to 25 cm²
  * wound hematoma greater than or equal to 100 cm²
  * spontaneous nose bleed lasting longer than 5 min
  * macroscopic hematuria spontaneous or lasting longer than 24 hours if associated with an intervention
  * spontaneous rectal bleeding (more than a spot on toilet paper)
  * gingival bleeding lasting longer than 5 min
  * any other bleeding event considered clinically relevant by the investigator
  Minor bleeding events were defined as all other bleeding events that did not fulfil the criteria from above.
Time Frame: First administration until 12-15 days
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 857 | 871 | 868
Participants
  Major | 5 | 5 | 12
  Clinically relevant | 23 | 22 | 21
  Minor | 46 | 45 | 51
  None | 783 | 799 | 784
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.1416, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.0942, Fisher Exact

ADVERSE EVENTS:
Time Frame: First administration until (usually) day 21, i.e., treatment period + 3 days.
Description: Treatment emergent events (last medication + 3 days); The usual treatment period was 12 to 15 days with up to 18 days. Only one patient was treated for 33 days.
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Serious Adverse Events (participants affected / at risk) | 59/857 | 57/871 | 45/868
Other Adverse Events (participants affected / at risk) | 718/857 | 724/871 | 711/868
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 220mg (N=857) | Dabigatran 150mg (N=871) | Enoxaparin (N=868)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 2 | 4
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 5 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 5 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 0
Gait disturbance (General disorders) | 1 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 2 | 1
Pyrexia (General disorders) | 0 | 3 | 2
Secretion discharge (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1
Blister infected (Infections and infestations) | 1 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 3 | 2
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 2 | 3
Heart rate irregular (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Occult blood (Investigations) | 0 | 1 | 0
Occult blood positive (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Complex regional pain syndrome (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 2 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 10 | 9 | 5
Haematoma (Vascular disorders) | 2 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1 | 0
Vasospasm (Vascular disorders) | 0 | 1 | 0
Venous insufficiency (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 220mg (N=857) | Dabigatran 150mg (N=871) | Enoxaparin (N=868)
Anaemia (Blood and lymphatic system disorders) | 48 | 47 | 46
Constipation (Gastrointestinal disorders) | 229 | 268 | 245
Dyspepsia (Gastrointestinal disorders) | 41 | 39 | 44
Nausea (Gastrointestinal disorders) | 198 | 204 | 189
Vomiting (Gastrointestinal disorders) | 105 | 110 | 95
Oedema peripheral (General disorders) | 244 | 275 | 254
Pyrexia (General disorders) | 154 | 157 | 167
Anaemia postoperative (Injury, poisoning and procedural complications) | 48 | 63 | 64
Post procedural oedema (Injury, poisoning and procedural complications) | 60 | 61 | 52
Post procedural pain (Injury, poisoning and procedural complications) | 110 | 114 | 84
Body temperature increased (Investigations) | 48 | 58 | 60
Hypokalaemia (Metabolism and nutrition disorders) | 47 | 46 | 47
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 54 | 52
Joint swelling (Musculoskeletal and connective tissue disorders) | 40 | 35 | 44
Pain in extremity (Musculoskeletal and connective tissue disorders) | 55 | 69 | 67
Dizziness (Nervous system disorders) | 56 | 59 | 79
Headache (Nervous system disorders) | 36 | 46 | 37
Insomnia (Psychiatric disorders) | 100 | 105 | 109
Urinary retention (Renal and urinary disorders) | 72 | 82 | 60
Pruritus (Skin and subcutaneous tissue disorders) | 38 | 44 | 52
Deep vein thrombosis (Vascular disorders) | 86 | 93 | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract